CLINICAL TRIAL: NCT04393532
Title: Laparoscopic Primary Umbilical Hernia Repair With Routine Defect Closure Using Su2ura Approximation Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anchora Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANC-001
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Primary Umbilical Hernia
Keywords: hernia; umbilical; repair; primary; laparoscopic
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Intervention Model Description: All recruited patients will undergo a laparoscopic hernia repair procedure using the Su2ura Approximation Device.
Masking Description: single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic hernia repair using Su2ura Approximation Device (Experimental): Surgery will be performed under general anesthesia. Standard antibiotic prophylaxis will be administered at induction of anesthesia. A single surgeon, the PI, will perform the procedure. A surgical assistant will be selected by the PI from the surgical staff of the department.
  The procedure will involve placement of laparoscopic ports, reduction of the hernia sac, closure of the defect with the Su2ura Approximation device and fixation of mesh with tacks over the closed defect.
  Study follow up visits: at post operation discharge, 14 days, 3 months, 6 months.
  Interventions: Device: Su2ura Approximation Device; Procedure: Laparoscopic hernia repair surgery

INTERVENTIONS:
Device: Su2ura Approximation Device — the use of the study device during a laparoscopic surgery
Procedure: Laparoscopic hernia repair surgery — repairing primary umbilical hernia in a laparoscopic procedure using the study device.

SUMMARY:
Intended Use The Su2ura™ Approximation Device is indicated for tissue approximation in endoscopic and open surgery for the placement of interrupted or running stitches in soft tissue such as hernia repair

Objectives To assess the safety and efficacy of the Su2ura approximation device for the laparoscopic repair of primary umbilical hernia

Number of Subjects 45 patients

Number of Centers Two study centers in Israel and one in Slovenia.

Study Duration 6 months

Study Procedures Surgery will be performed under general anesthesia. Standard antibiotic prophylaxis will be administered at induction of anesthesia. A single surgeon, the PI, will perform the procedure. A surgical assistant will be selected by the PI from the surgical staff of the department.

The procedure will involve placement of laparoscopic ports, reduction of the hernia sac, closure of the defect with the Su2ura approximation device and fixation of mesh with tacks over the closed defect.

Study follow up visits: at post operation discharge, 14 days, 3 months, 6 months.

Study follow up procedures:

Also include SAE's and SADE's during follow up

1. Quality of life questionnaire: patient-reported satisfaction and function will be assessed through the validated, hernia-specific European Hernia Society Quality of Life questionnaire (EuraHS-QoL)
2. Clinical testing to determine hernia recurrence and clinical bulging

Statistical analysis The sample size calculation based on the Exact Binomial distribution. The investigators will compute the 95% confidence intervals for a binomial probability, relying on the Clopper-Pearson (exact) method.

DETAILED DESCRIPTION:
DEVICE NAME AND INTENDED USE Device Name Su2ura™ Approximation Device

Intended Use The Su2ura™ Approximation Device ("Su2ura approximation device") is indicated for tissue approximation in endoscopic surgery for the placement of interrupted or running stitches in soft tissue such as hernia repair.

DEVICE DESCRIPTION Su2ura™ Approximation Device is a manual tissue approximation device comprised of an ergonomic Handle and Anchors threaded with suture.

Device Operation When using the Su2ura Approximation Device for suturing and approximation in MIS, the device is inserted through a 5mm port into the abdominal cavity and placed against the tissue. The surgeon presses the trigger to deploy threaded anchors into the tissue. Each anchor with a suture is placed with one single action. The surgeon may repeat the deployment operation several times at different target sites, as needed to form a short/long interrupted or running stitch. The device User Manual includes a recommendation to perform 4 continuous anchors each time whereas this process can be repeated again and again until the area is fully sutured. For approximation of the tissue after the anchors are positioned, the surgeon retracts the device from the port and ties an extracorporeal unidirectional surgical knot. The surgeon then changes the toggle into tightening mode and mounts the Cap on the shaft. The surgeon re-inserts the shaft through the port and slides the knot towards the approximation site using the tightening knob to collect thread and approximating the incision edges. The surgeon uses laparoscopic scissors to cut the thread and may repeat the suturing process again several times as needed until the incision is fully closed.

RISKS and BENEFITS The su2ura approximation device is designed according to international standards for medical devices. Compliance with these standards ensures that the device can be used safely in human beings.

Biocompatible materials are used for the device components. The use of biocompatible materials should protect the subject from hazardous adverse events.

Risks

The following general risks/complications may be related to the use of Su2ura Approximation Device:

* Pain due to tissue penetration or approximation
* Vessel/nerve injury during insertion
* Su2ura approximation device migration
* Adhesions The Su2ura Approximation Device was subjected to a series of pre-clinical tests in order to verify its safety and usability. In addition, the device is restricted for use by a trained physician, and all relevant warnings and precautions are clearly indicated in the Instructions for Use document (Version 1.0) of the device. The full Risk Analysis is described in "Risk Management" of Su2ura Approximation Device Version 1.0.

Risk Mitigation Risk analysis is performed according to the standard ISO 14971 Medical Device Risk Analysis. Potential electrical, mechanical and biological hazards are identified, risks are evaluated, risk mitigation is implemented and verified.

Benefits Laparoscopic hernia repair, due to its clinical benefits of quick recovery, fewer complications and low recurrence rate, has become a favorable and standard technique.

In open hernia surgery, the standard procedure includes reapproximation of the fascia in the midline and restoration of the abdominal wall, followed by application of surgical mesh.

This reapproximation of fascia in the midline is more complex in laparoscopic hernia repair; therefore, this has not become standard practice4. Laparoscopic repair typically concludes with mesh placement bridging over open defects, with no sutured defect closure5. The bridging technique without defect closure results in higher rate of recurrence. When the defect is sutured at laparoscopy, clinical studies show a significant reduction in recurrence rates4.

Notwithstanding the above mentioned, it is important to note that whether or not primary closure of the defect is performed in both open and laparoscopic hernia surgery, the use of surgical mesh is essential and has become standard, with a lower incidence of recurrence6.

For laparoscopic fixation of the mesh, several techniques are available, where the most frequent involve intra-abdominal fixation with sutures or tackers (staples) or transabdominal suture fixation. Complications related to the use of transabdominal suturing or stapling include mesh migration or folding, infection, post-operative pain and recurrence4.

Therefore, there is a need for novel devices to: a) enable primary intra-abdominal defect closure during laparoscopic surgery; b) provide a simple and safe alternative to transfascial suture fixation of surgical mesh; and, c) standardize a technique for defect closure and for surgical mesh fixation in laparoscopic procedures.

STUDY OBJECTIVE The objectives are to assess the safety and efficacy of the Su2ura approximation device for the laparoscopic repair of primary umbilical hernia.

Duration of Study Study duration includes a minimum hospitalization period of 1 to 2 days, followed by patient visits at 14 days, 3 months, 6 months after surgery.

The actual point of enrollment of the subject is considered the day of the surgery.

STUDY TREATMENT Study Design The study is a prospective, triple -center, two countries, open study to evaluate the efficacy and safety of the su2ura approximation device.

The study will be performed in the Department of Surgery at Ziv Medical Center, Safed, Israel, Department of Surgery at Barzilai Medical Center, Ashkelon, Israel and at the Surgery Department of General Hospital Izola, Polje 40, 6310 Izola, Slovenia Data reporting will be done on a Case Report Form (eCRF). Eligible patients with a primary umbilical hernia, desiring elective surgical repair and meeting the inclusion criteria will be offered participation in this study. The background of the proposed study and the risks and benefits will be explained to the patient, informed consent taken and the study consent form signed.

The study subject will be invited for 8 visits: Screening, Baseline, post-operative discharge, and at 14 days, 3 months, 6 months after surgery.

During the visits, an interview will be conducted, where the following topics will be discussed: the occurrence of adverse events, compliance in the reporting of adverse events and an update on concomitant medication.

Data collection will include physician identification, investigational device identification data and usage of the device. This data will be documented on the CRF, together with the occurrence of any adverse events during device usage.

All adverse events reported by study subjects (whether device related or not) will be recorded during the course of the clinical study. All serious adverse events/complications will be reported immediately (within 24 hours) to the study sponsor/monitor, the Institutional Review Board and in accordance with local regulatory requirements.

Medical History The following demographic and medical information from the subject and the subject's medical chart will be recorded: age; gender; weight; height; body mass index (BMI), number of births, previous medical history and co-morbidities; list of concomitant medication; and, smoking history.

The information will be recorded in the CRF for all subjects participating in this study.

Hernia History Full history of the umbilical hernia will be recorded on the CRF, including information on symptoms, duration, previous treatment, and a list of concomitant medication.

Physical Examination During the screening visit all subjects will undergo a standard physical examination by an authorized physician. The physician's evaluation will include diagnosis and documentation of any significant clinical abnormality or disease.

Blood and urine tests During the screening visit all subjects will undergo hematology and biochemistry blood tests.

Blood hematology test will include a CBC and blood chemistry test will include the following measures: Sodium (Na), Potassium (K), Chloride (Cl), Creatinine, Glucose, Urea, Albumin, Calcium total, Alkaline Phosphatase (ALP), ALT, AST, Total Bilirubin, Direct Bilirubin, LDH, Total Protein, Uric Acid, CRP, and Lipid Profile (including Total Cholesterol, HDL, LDL, Triglycerides.

Urine pregnancy test will be performed during the screening visit.

Screening visit (day -7) Subjects will be asked to sign a consent form and will be screened for study eligibility according to inclusion and exclusion criteria. The hernia will be thoroughly assessed. Subject demographic and medical information acquired from the subject or the subject's medical chart, including age, gender, previous medical history, concomitant medications, risk factors etc. will be also recorded on the CRF.

In addition, subjects will undergo a physical examination, vital sign measurements and blood tests. Quality of life questionnaire: patient-reported satisfaction and function will be assessed through the validated, hernia-specific European Hernia Society Quality of life questionnaire (EuraHS-QoL).

The investigator will confirm their eligibility and their physical and mental suitability to participate in this study.

Baseline visit, Surgery (day 0) The baseline visit is the stage at which surgery is performed. Patients will already have been assessed 2 or 3 weeks earlier in the preassessment clinic where fitness for surgery is verified and clinical investigation or treatment for optimization for surgery organized. Thereafter, patients will be admitted to the Department of Surgery at Ziv Medical Center either on the morning of surgery or the day prior to surgery for final preoperative preparation. Surgery in all cases will be laparoscopic umbilical hernia repair. No other elective surgical procedure will be performed during the same visit.

Surgery will be performed under general anesthesia. Standard antibiotic prophylaxis will be administered at induction of anesthesia. A single surgeon, the PI, will perform the procedure. A surgical assistant will be selected by the PI from the surgical staff of the department.

Patients will be placed in the supine position. Standard skin preparation with povidone iodine solution will be performed. A 12 to 14 mm Hg carbon dioxide pneumoperitoneum will be achieved using a Verres needle and maintained throughout surgery. Three laparoscopic ports will be inserted: the first, a 5mm port in the left anterior axillary line 2 cm below the costal margin; the second, a 10 mm port at the level of the umbilicus or in the transcrestal plane; the third, a 5mm port 2 cm below the line of the second port. A 5 or 10 mmm 30 degree camera will be connected to an Olympus or Storz Medical Systems video laparoscopic stack. The video of the surgical procedure will be recorded and stored with the CRF.

The umbilical hernia will be visualized (any adhesions at or close to the area of repair will be divided). At the time of surgery the hernia sac is most likely sac will be dissected free already; if not, the sac will be dissected free of the defect at the umbilicus - the sac and hernia then drops into the abdominal cavity. The abdominal contents will be inspected. The hernia defect will be inspected and the Su2ura approximation device will then be used to close the defect, placing stainless steel implantable anchors threaded on a Polyethylene braided surgical suture no less than 5mm and no more than 15 mm apart. After the approximation, the sutures will be locked with extracorporeal knot. Mesh will be placed according to the guidelines and the clinical status. After one last check of hemostasis and the integrity of the repair, the laparoscopic ports and instruments will be withdrawn under vision, and the pneumoperitoneum released.

Postoperatively, the patient will be transferred to the recovery area and then the surgical ward, where the patient will be monitored by the medical and nursing staff of the Department of Surgery. It is expected that the patients will spend one postoperative night in the department and be discharged the following day.

Pain medication prescribed will be at the discretion of the anesthesiologist during and immediately after surgery. In the Department of Surgery, patients will be prescribed standard oral pain medication (usually metamizole - Optalgin - unless a contraindication exists) to continue after discharge, and receive standard advice on physiotherapy, mobility, and the resumption of physical activity and work.Follow up visits (day 14 (± 2days), 3 months (± 1 week), 6 months (± 1 week) During the follow up visits, subjects will undergo physical examination, vital sign measurements and blood tests. Information on adverse events and concomitant medications will be collected.

Study follow up procedures will be performed:

1. Quality of life questionnaire: patient-reported satisfaction and function will be assessed using the validated, hernia-specific European Hernia Society quality of life questionnaire (EuraHS-QoL)
2. Clinical examination to determine the presence of hernia recurrence and clinical bulge
3. SAE's SADE's Seroma

Concomitant medication All medication taken by the subject is termed 'concomitant' medication. All concomitant medication taken during the study must be documented in the case report form (name of drug, date drug started, dosage, number of times drug taken daily, route of medication, and indication for prescription).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient desires elective surgical repair
* Patient is able to give informed consent
* Diagnosis of a primary umbilical hernia with a fascial defect of width no more than 5 cm in size on clinical examination or CT scan
* Body mass index (BMI) 20-40 kg/m2
* Candidate for laparoscopic repair based on the operating surgeon's assessment

Exclusion Criteria:

* Non-primary or incisional hernia in the umbilical hernia
* Diagnosis of concomitant abdominal wall defect(s) contiguous with primary umbilical hernia
* Patient previously underwent open or laparoscopic umbilical hernia repair surgery
* Patient previously underwent open or laparoscopic abdominal surgery which spans the umbilical area
* Patient in need of concomitant non-hernia repair surgical procedure(s)
* Patient in need of emergent primary umbilical hernia repair for complications such as incarceration, intestinal obstruction or strangulation
* The patient desires hernia repair using a technique other than that consistent with the study
* Patient has loss of domain as assessed on physical examination or CT scan
* Patient has a severe co-morbid condition likely to limit survival to less than 2 years
* Patient was treated with chemotherapy in the past 6 months
* Patient was treated with steroids in the past 6 months
* Pre-operative or intra-operative contamination of the surgical site
* Patient with known collagen disorder
* Patient is pregnant or intends to become pregnant during the study period
* Patient has ascites on physical examination or CT scan
* Patient has cirrhosis
* Patient undergoing dialysis treatment
* Patient has a wound-healing disorder
* Patient has an untreated coagulation disorder or is on anti-coagulant therapy not managed peri-operatively with the advice or supervision of a hematologist
* Patient with autoimmune disorder requiring more than 10 mg of corticosteroid daily
* Patient who is immunocompromised (including a diagnosis of HIV/AIDS, organ transplant, or receiving chemo- or radiation therapy
* Non-compliance with the study protocol
* Patient requests to exist the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Overall rate of Serious Adverse Events and serious adverse device effects (SADE) up to hospital discharge and up to the 60th post-operative day. | 60 days from baseline
  AEs and SADEs will be documented and reviewed to assess the safety of the device

SECONDARY OUTCOMES:
Hernia Recurrence Rate at 6 months (Investigator confirmed hernia recurrence on physical examination) | 6 months
  During follow-up period patients with reaccuring hernia will be documented and reviewed to assess the efficacy of this device
Patient satisfaction and function as assessed by the European Hernia Society quality of life questionnaire (EuraHS-QoL) at a 6-month follow up. Score range : 0-180, lower score indicates less pain and discomfort. | 6 months
  During follow-up period patients satisfaction will be followed and documented and reviewed to assess the efficacy of this device
Clinical bulging defined as any bulge of tissue or mesh beyond the natural contour of the abdomen on supine flexion at 6 months follow up. | 6 months
  During follow-up period patients with tissue bulging will be documented and reviewed to assess the efficacy of this device
Evidence of seroma defined by clinical examination up to 6 months after surgery | 6 months
  During follow-up period patients with seroma will be documented and reviewed to assess the efficacy of this device

CONTACTS AND LOCATIONS:
Overall Officials: Yoni Epstein, Study Director — Anchora Medical
Locations (3):
- Israel (2):
  - Ziv Medical Center, Safed, North
  - Barzilai Medical Center, Ashkelon, South
- Splošna bolnišnica Izola (General Hospital Izola), Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bittner R, Bingener-Casey J, Dietz U, Fabian M, Ferzli GS, Fortelny RH, Kockerling F, Kukleta J, Leblanc K, Lomanto D, Misra MC, Bansal VK, Morales-Conde S, Ramshaw B, Reinpold W, Rim S, Rohr M, Schrittwieser R, Simon T, Smietanski M, Stechemesser B, Timoney M, Chowbey P; International Endohernia Society (IEHS). Guidelines for laparoscopic treatment of ventral and incisional abdominal wall hernias (International Endohernia Society (IEHS)-part 1. Surg Endosc. 2014 Jan;28(1):2-29. doi: 10.1007/s00464-013-3170-6. Epub 2013 Oct 11. PMID 24114513
- [Background] Baylon K, Rodriguez-Camarillo P, Elias-Zuniga A, Diaz-Elizondo JA, Gilkerson R, Lozano K. Past, Present and Future of Surgical Meshes: A Review. Membranes (Basel). 2017 Aug 22;7(3):47. doi: 10.3390/membranes7030047. PMID 28829367
- [Background] Zendejas B, Hernandez-Irizarry R, Ramirez T, Lohse CM, Grossardt BR, Farley DR. Relationship between body mass index and the incidence of inguinal hernia repairs: a population-based study in Olmsted County, MN. Hernia. 2014 Apr;18(2):283-8. doi: 10.1007/s10029-013-1185-5. PMID 24233340
- [Background] Franz MG. The biology of hernia formation. Surg Clin North Am. 2008 Feb;88(1):1-15, vii. doi: 10.1016/j.suc.2007.10.007. PMID 18267158
- [Background] Dabbas N, Adams K, Pearson K, Royle G. Frequency of abdominal wall hernias: is classical teaching out of date? JRSM Short Rep. 2011 Jan 19;2(1):5. doi: 10.1258/shorts.2010.010071. PMID 21286228
- [Background] Umbilical Hernia. Anouchka H. Coste; John D. Parmely. Jan 2019
- [Background] Yuri W. Novitsky. Hernia Surgery, Current Principles (Page 231)
- [Background] Hjaltason E. Incarcerated hernia. Acta Chir Scand. 1981;147(4):263-7. PMID 7324753
- [Background] Kaufmann R, Halm JA, Eker HH, Klitsie PJ, Nieuwenhuizen J, van Geldere D, Simons MP, van der Harst E, van 't Riet M, van der Holt B, Kleinrensink GJ, Jeekel J, Lange JF. Mesh versus suture repair of umbilical hernia in adults: a randomised, double-blind, controlled, multicentre trial. Lancet. 2018 Mar 3;391(10123):860-869. doi: 10.1016/S0140-6736(18)30298-8. Epub 2018 Feb 17. PMID 29459021
- [Background] Zeichen MS, Lujan HJ, Mata WN, Maciel VH, Lee D, Jorge I, Plasencia G, Gomez E, Hernandez AM. Closure versus non-closure of hernia defect during laparoscopic ventral hernia repair with mesh. Hernia. 2013 Oct;17(5):589-96. doi: 10.1007/s10029-013-1115-6. Epub 2013 Jun 20. PMID 23784711
- [Background] Bittner R, Bingener-Casey J, Dietz U, Fabian M, Ferzli G, Fortelny R, Kockerling F, Kukleta J, LeBlanc K, Lomanto D, Misra M, Morales-Conde S, Ramshaw B, Reinpold W, Rim S, Rohr M, Schrittwieser R, Simon T, Smietanski M, Stechemesser B, Timoney M, Chowbey P. Guidelines for laparoscopic treatment of ventral and incisional abdominal wall hernias (International Endohernia Society [IEHS])-Part III. Surg Endosc. 2014 Feb;28(2):380-404. doi: 10.1007/s00464-013-3172-4. Epub 2013 Sep 17. No abstract available. PMID 24043642
- [Background] Wright BE, Beckerman J, Cohen M, Cumming JK, Rodriguez JL. Is laparoscopic umbilical hernia repair with mesh a reasonable alternative to conventional repair? Am J Surg. 2002 Dec;184(6):505-8; discussion 508-9. doi: 10.1016/s0002-9610(02)01071-1. PMID 12488148
- [Background] Olsen MA, Nickel KB, Wallace AE, Mines D, Fraser VJ, Warren DK. Stratification of surgical site infection by operative factors and comparison of infection rates after hernia repair. Infect Control Hosp Epidemiol. 2015 Mar;36(3):329-35. doi: 10.1017/ice.2014.44. PMID 25695175
- [Background] Heniford BT, Park A, Ramshaw BJ, Voeller G. Laparoscopic repair of ventral hernias: nine years' experience with 850 consecutive hernias. Ann Surg. 2003 Sep;238(3):391-9; discussion 399-400. doi: 10.1097/01.sla.0000086662.49499.ab. PMID 14501505
- [Background] Rutkow IM. Demographic and socioeconomic aspects of hernia repair in the United States in 2003. Surg Clin North Am. 2003 Oct;83(5):1045-51, v-vi. doi: 10.1016/S0039-6109(03)00132-4. PMID 14533902
- [Background] Aguirre DA, Santosa AC, Casola G, Sirlin CB. Abdominal wall hernias: imaging features, complications, and diagnostic pitfalls at multi-detector row CT. Radiographics. 2005 Nov-Dec;25(6):1501-20. doi: 10.1148/rg.256055018. PMID 16284131